CLINICAL TRIAL: NCT04388228
Title: Audit and Feedback for General Practitioners in the Intego Network
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study is not applicable anymore due to the Covid pandemic.
Sponsor: Tine De Burghraeve (Other)
Responsible Party: Sponsor-Investigator, Tine De Burghraeve, Tine De Burghraeve, PhD, KU Leuven
Organization: KU Leuven (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: S62753
Record Dates: First submitted 2020-05-11; First posted 2020-05-14 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Diabetes Mellitus; Chronic Kidney Diseases; Heart Failure
MeSH Terms: conditions — Diabetes Mellitus; Renal Insufficiency, Chronic; Heart Failure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Extended audit and feedback (Experimental): The intervention consists of an extended electronically delivered feedback with multiple components which will be delivered 4 times electronically into general practices over 12 months.
  This extended feedback report consists of:
  * Benchmarking of the results of the audit versus peers, versus guidelines and versus disease specific laboratory results.
  * A low cognitive load of the feedback where the results will be presented with the help of graphs.
  * Action plans to improve the quality of registration
  * A push system to minimize the effort the GP must make to consult the feedback.
  Interventions: Other: Extended audit and feedback in GPs electronic health record
- Basic feedback (Active Comparator): In the past, all GPs received basic feedback on the level of registration in the EHR and this form of feedback will still be provided in the control group. By providing all GPs a basic level of feedback, we do not change the former protocol and all GPs will receive the opportunity to improve their registration performance. Only the way of receiving feedback is more straightforward, the GP needs to login to HealthStat.be.
  Interventions: Other: Extended audit and feedback in GPs electronic health record

INTERVENTIONS:
Other: Extended audit and feedback in GPs electronic health record — The intervention consists of an extended electronically delivered feedback with multiple components which will be delivered 4 times electronically into general practices over 12 months.
  This extended feedback report consists of:
  * Benchmarking of the results of the audit versus peers, versus guidelines and versus disease specific laboratory results.
  * A low cognitive load of the feedback where the results will be presented with the help of graphs.
  * Action plans to improve the quality of registration
  * A push system to minimize the effort the GP must make to consult the feedback.

SUMMARY:
Audit and feedback is an extensively investigated quality intervention, which according to the last Cochrane review leads to small but potentially important improvements in professional practice. There is some evidence that feedback can improve EHR registration but the effect and important features of feedback are still the subject of debate. Previous work has identified some testable and theory-informed hypotheses for designing an audit and feedback intervention and suggestions to improve the effectiveness of the intervention are available in literature. There are several criteria feedback could meet to have an impact on the registration level of GP's in the EHR. The researchers now want to evaluate if the effort to make an extended feedback intervention has an effect on the registration behavior of the GP.

The research question is: Does an audit and extended feedback intervention improves the quality of registration in the EHR of the general physician compared to basic feedback?

DETAILED DESCRIPTION:
Intego is a Belgian general practice-based morbidity registration network at the Department of General Practice of the University of Leuven. Intego collects data on health parameters, incidence and prevalence rates, laboratory results, and prescribed drugs for all relevant subgroups. It is unique in Belgium. These data are used as a basis for teaching, quality improvement interventions, and research, as well as for policy making by both physicians' organizations and governmental bodies. The health ministry of the Flemish government mainly funds the network. Ad hoc research projects serve as an additional funding source.

Up until 2017, 97 general practitioners (GP's) of 55 practices evenly spread throughout Flanders, Belgium, collaborated in Intego. GP's applied for inclusion in the registry. Before acceptance of their data, registration performance was audited using algorithms to compare their results with those of all other applicants. Only data of practices with optimal registration performance that met our three quality requirements were included in the database. First, the average number of new diagnoses per patient per year should be higher than one. Second, diagnoses have to be entered in the practice software using keywords. The Intego GP's prospectively and routinely registered all new diagnoses and new drug prescriptions, as well as laboratory test results and patient information. The registration made use of computer-generated keywords internally linked to codes [International Classification of Primary Care (ICPC-2) and International Statistical Classification of Diseases and Related Health Problems 10th Revision (ICD-10) for diagnoses and WHO's Anatomical Therapeutic Chemical (ATC) classification system for drugs]. The percentage of diagnoses recorded without using keywords should be less than 5%. Finally, these parameters must remain stable for at least three years.

In 2017, Intego made a transition in data infrastructure and size of the network.

Further information technology development for the electronic health record (EHR) 'Medidoc' was terminated, and all its users were urged by the vendor to migrate to a new EHR, called CareConnect (Corilus), a cloud-based EHR. This transition marked the moment to redesign the data collection for this registry, which had not changed since its start. To comply with the new General Data Protection Regulation legislation, the Healthdata.be platform was identified as a partner for this task.

Moreover, the number of practices was increased and now counts 107 practices (410 GPs). However, new GP practices might not meet the quality requirements for good registration yet.

The data completeness of the EHR is thus an important factor to consider when reusing data stored in the EHR. Other pitfalls and sources of bias when using EHR data have also been identified. In order to improve registration, we want to implement extended electronically delivered feedback and evaluate its effects on correctly registering the diagnosis of chronic diseases and lifestyle habits in the EHR.

Audit and feedback is an extensively investigated quality intervention, which according to the last Cochrane review leads to small but potentially important improvements in professional practice. There is some evidence that feedback can improve EHR registration but the effect and important features of feedback are still the subject of debate. Previous work has identified some testable and theory-informed hypotheses for designing an audit and feedback intervention and suggestions to improve the effectiveness of the intervention are available in literature. There are several criteria feedback could meet to have an impact on the registration level of GP's in the EHR. We now want to evaluate if the effort to make an extended feedback intervention has an effect on the registration behavior of the GP.

The research question is: Does an audit and extended feedback intervention improves the quality of registration in the EHR of the general physician compared to basic feedback?

ELIGIBILITY:
inclusion criteria:

* This trial has the general practices as the level of allocation.
* All GPs in the Intego network will be asked to participate in this trial.
* For GPs working in a group, the whole group will be asked to collaborate.

Exclusion criteria:

- If not all GPs in a group practice want to collaborate in the intervention study, the whole GP practice will not be included in this study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01-30 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
percentage registered diagnoses of DM 2 in the EHR | 12 months
  Registered diagnosis of type II diabetes in GPs electronic health record

SECONDARY OUTCOMES:
Percentage registered lifestyle factors | 12 months
  Registration of lifestyle habits such as alcohol and tobacco use
percentage registered diagnoses of heart failure | 12 months
  Registered diagnosis of heart failure in GPs electronic health record

OTHER OUTCOMES:
CKD follow-up quality indicator | 12 months
  Percentage of patients with CKD in whom the GFR, albuminuria and total protein is determined at least once a year
CKD vaccination quality indicator | 12 months
  Percentage of patients with CKD who received a pneumococcal vaccination
Diabetes treatment quality indicator | 12 months
  Percentage of patients with diabetes and CKD who no longer receive metformin
Diabetes follow-up quality indicator | 12 months
  Percentage of patients with diabetes whose HbA1c level is measured at least once every 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Tine De Burghgraeve, PhD, Principal Investigator — KU Leuven

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Van den Bulck S, De Burghgraeve T, Raat W, Mamouris P, Coursier P, Vankrunkelsven P, Goderis G, Hermens R, Van Pottelbergh G, Vaes B. The effect of automated audit and feedback on data completeness in the electronic health record of the general physician: protocol for a cluster randomized controlled trial. Trials. 2021 May 4;22(1):325. doi: 10.1186/s13063-021-05259-9. PMID 33947448